CLINICAL TRIAL: NCT06203834
Title: Evaluating the Efficacy of I-fiber Pearl on Reducing Body Fat Accumulation in Obese Subjects: a Randomized, Double-blind, and Placebo-controlled Trial
Brief Title: Evaluating the Efficacy of I-fiber Pearl on Reducing Body Fat Accumulation in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Collaborators: ITSWAY BIOTECH INC. (Unknown)
Responsible Party: Principal Investigator, Chin-Lin Hsu, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CS2-23093
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- placebo (Placebo Comparator): Placebo 200g, without any ingredients of inulin fiber. Eat 200g for once, and once a day.
  Interventions: Dietary Supplement: placebo
- I-Fiber Pearl (Experimental): I-Fiber Pearl 200g, with inulin fiber. Eat 200g for once, and once a day.
  Interventions: Dietary Supplement: I-Fiber Pearl

INTERVENTIONS:
Dietary Supplement: I-Fiber Pearl — Eat 200g for once, and once a day.
  Arms: I-Fiber Pearl
Dietary Supplement: placebo — Eat 200g for once, and once a day.
  Arms: placebo

SUMMARY:
The aim of this study is to investigate the effects of I-Fiber Pearl on Body Weight and Body Fat in Obese Adults.

DETAILED DESCRIPTION:
This randomized, double-blinded,placebo-controlled clinical trial will be conduct for 12 weeks with fifty adults. Subjects will be recruited and randomly assigned into two groups: (1) placebo, n = 25; (2) I-Fiber Pearl, n=25. During the 12 weeks intervention, the subjects should take 200g placebo or 200g I-Fiber Pearl a day . The two pearl are supplied in plastic packages, and both the products taste the same. Subjects also should complete the assessment of anthropometric measurement, intestinal questionnaire , food record, urine, feces and blood collection at week 0 and week 12.

ELIGIBILITY:
Inclusion Criteria:

* female
* aged 20-50 years old
* body mass index is greater than or equal to 27 kg/m2
* waist greater than or equal to 80 cm

Exclusion Criteria:

* Subjects diagnosed with cancer and on curative care.
* Subjects diagnosed with heart disease and on curative care.
* Subjects who use other drugs whose pharmacological effects may affect the experiment or may aggravate the effects of the drug.
* Subjects with systemic infection requiring antibiotics.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Change from baseline body weight at week 12 | Week 0, Week 12
  Compared the difference of body weight between the week 12 and 0.
Change from baseline body fat at week 12 | Week 0, Week 12
  Compared the difference of body fat between the week 12 and 0.

CONTACTS AND LOCATIONS:
Overall Officials: Chin-Lin Hsu, Ph.D., Study Chair — Chung Shan Medical University; Chin-Lin Hsu, Ph.D., Principal Investigator — Chung Shan Medical University; Shiuan-Chih Chen, Dr., Principal Investigator — Chung Shan Medical University; Hung-Hsuan Kuo, Master, Principal Investigator — Chung Shan Medical University; Chun-Tse Tsai, Master, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, South, Taiwan